CLINICAL TRIAL: NCT02011451
Title: Safety and Neuroprotective Effects of Theaphenon 95% (95% Pure EGCG) in Multiple Sclerosis
Brief Title: Safety and Brain Protection Effects of the Green Tea Extract Theaphenon 95% (95% Pure EGCG) in Multiple Sclerosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: unable to enroll
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Jesus Lovera MD, Assistant Professor, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4818-A-1; 4816-A-1 (Other Grant/Funding Number: National MS Society)
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Green Tea; ECGC; Theaphenon; Randomized placebo controlled trial; NAA; Spectroscopy; Brain Atrophy; SIENA
MeSH Terms: conditions — Multiple Sclerosis | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 95% Pure ECGC capsules 200mg (Experimental): 95% Pure ECGC capsules 200mg three times a day with food for 6 months
  Interventions: Drug: 95% Pure ECGC capsules 200mg
- Sugar pill (Placebo Comparator): Matched placebo capsules
  Interventions: Drug: Placebo Comparator:

INTERVENTIONS:
Drug: 95% Pure ECGC capsules 200mg — Theaphenon 95% 95% Pure EGCG
  Other Names: Theaphenon 95%
  Arms: 95% Pure ECGC capsules 200mg
Drug: Placebo Comparator:
  Other Names: "Sugar pill"
  Arms: Sugar pill

SUMMARY:
The hypothesis is that 95% pure EGCG can protect brain cells in patients with Multiple Sclerosis. To test this hypothesis we are going to compare the changes in n-Acetyl-Aspartate (a chemical that reflects the number of neurons and their metabolism) over one six between people with MS treated with EGCG at a dose of 400mg twice a day and people with MS treated with a matching sugar pill.

DETAILED DESCRIPTION:
This will be a double blind placebo controlled trial of Theaphenon 95% (95% pure Epigallo-catechin-galleate [EGCG]) as a treatment for MS.

The primary outcome will be the changes in N-Acety-Aspartate (NAA) levels over six months. Secondary outcomes will be changes in brain atrophy over over six months. As an exploratory outcome we will correlate changes in NAA levels with free Plasma levels of EGCG 8 hours after the morning dose.

Exploratory outcomes include disability progression by Expanded Disability Status Scale (EDSS), multiple sclerosis functional composite components and a cognitive test battery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS by McDonald criteria
* Relapsing-remitting MS or secondary progressive MS
* Stable therapy with Copaxone, Rebif, Betaseron or Avonex 30 mcg for at least six months
* EDSS Score less than or equal to 7.0
* Ages 18-60.
* Participants must have normal organ and marrow function as defined below:

  * Leukocytes ≥3,000/µL
  * Absolute neutrophil count ≥1,500/µL
  * Platelets ≥100,000/µL
  * Total bilirubin ≤local upper limit of normal
  * AST (SGOT) ≤local upper limit of normal
  * ALT (SGPT) ≤local upper limit of normal
  * Creatinine ≤local upper limit of normal

Exclusion Criteria:

* MS relapse within the 30 days prior to enrollment
* A primary progressive form of MS.
* Previous treatment prior to study entry as follows: complete radiation ablation of the bone marrow or anti-CD4 antibody treatment (Campath) at any time; mitoxantrone, cyclophosphamide, Natalizumab or other immunomodulatory or immunosuppressant therapies except the DMT's included in the inclusion criteria and methylprednisone for relapses within prior nine months.
* History of renal or liver disease.
* Consumption of green tea or supplements containing green tea or tea extract within 30 days prior to enrollment.
* Participants may not participate in any other clinical trial involving investigational agents during the study, or within six months prior to enrolling in the study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Polyphenon E, tea, or any of the inactive ingredients present in the active or placebo capsules, including gelatin.
* History of allergic reactions to gadolinium or any other condition contraindicated for MRI.
* Uncontrolled, clinically-relevant active illness (aside from MS) including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any condition which would make the subject, in the opinion of the investigator, unsuitable for the study
* Inability to complete the baseline MRI scan
* Pregnant women
* Any underlying predisposition to gastrointestinal bleeding (peptic ulcer disease, gastritis, diverticulitis, colitis, hemorrhoids)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Rate of change in NAA levels adjusted for water content. | 6 months
  The rate of change will be calculated using all the time points available (baseline,3 and 6 months) using a mixed model analysis with the Log NAA as the dependent variable and water content, %grey matter, %white matter, %cerebrospinal fluid (CSF) and % lesion volume as covariates. All the voxels available for each subject where estimates have a standard deviation(SD) <30 will be used. A spatial anisotropic exponential covariance structure will be used.

SECONDARY OUTCOMES:
Brain Atrophy | 6 months
  Difference between the two groups in brain atrophy as measured by SIENA

CONTACTS AND LOCATIONS:
Locations (1):
- LSU Health Sciences Center, New Orleans, Louisiana, United States